CLINICAL TRIAL: NCT06291116
Title: Safety of RotigotiNe in Patients With Autosomal Dominant Polycystic Kidney Disease
Acronym: ETERNAL-PKD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/0345/HP
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental): Experimental group: standard care + rotigotine at 4 mg/24 hours for 24 months.
  Interventions: Drug: standard care + rotigotine at 4 mg/24h for 24 months.
- Control (Active Comparator): Control group: standard care for 24 months.
  Interventions: Drug: standard care for 24 months.

INTERVENTIONS:
Drug: standard care + rotigotine at 4 mg/24h for 24 months. — standard care + rotigotine at 4 mg/24h for 24 months.
  Arms: experimental
Drug: standard care for 24 months. — standard care for 24 months.
  Arms: Control

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is the most common hereditary kidney disease linked to mutation of the PKD1 or PKD2 genes encoding polycystins 1 and 2. Patients develop renal cysts with progressive impairment of renal function leading to renal failure. terminal renal failure for 1/3 of them. These patients also present early with high blood pressure and cardiovascular complications, notably intracerebral aneurysms. This phenotype is linked to abnormal polycystins on the cilia of renal epithelial and vascular endothelial cells which no longer ensure the mechanotransduction of shear forces linked to urinary and blood flow leading to the modification of numerous cellular functions.

Experimental results suggested that stimulation of dopamine receptor type 5 (DR5) could restore the mechanosensitivity of endothelial cells, a hypothesis supported by our first results showing that local administration of dopamine improves endothelial function in patients with ADPKD. through restoration of endothelial NO release upon increased blood flow. Similar positive results on endothelial function and hemodynamics were recently obtained in the IMPROVE-PKD study with rotigotine, a dopamine agonist administered via transdermal patches for 2 months at a low dose (4 mg/24h).

Dopaminergic stimulation could also prevent abnormalities linked to polycystin deficiency at the renal level and we therefore hypothesize that rotigotine could slow the progression of ADPKD both at the renal and cardiovascular levels.

This phase 2 study aims to ensure the good long-term tolerance of rotigotine in patients with ADPKD and to collect preliminary data on its renal impact.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients aged 18 to 60 years
* Normotensive or hypertensive patients treated controlled (SBP/DBP on daytime ABPM <135/85 mmHg less than 3 months old)
* Patient having read and understood the information letter and signed the consent form
* Effective contraception in women of childbearing age (for postmenopausal women, a confirmatory diagnosis should be obtained)
* Patient benefiting from a social protection scheme

Exclusion Criteria:

* Stage 4 or 5 renal insufficiency (GFR CKD-EPI <30 ml/min)
* Renal transplant patients
* Dialysis patients
* History of myocardial infarction or stroke less than 6 months old
* Severe hepatic insufficiency (Child-Pugh class C)
* Patients currently being treated or treated in the 6 months preceding the trial with a dopamine agonist or antagonist
* Systolic heart failure requiring hospitalization in the 6 months preceding inclusion or known heart failure with an LVEF <30%
* Orthostatic hypotension (decrease > 20 mm Hg)
* Pregnant, breastfeeding woman, or proven absence of contraception
* Excessive alcohol consumption (greater than 20 g/day)
* History of addictive behavior, particularly gambling, compulsive purchasing or hypersexuality
* Drug addiction or suspected illicit drug use
* Taking other sedative medications or other central nervous system depressants (benzodiazepines, antipsychotics, antidepressants or neuroleptics with antiemetic intent)
* Hypersensitivity to the active ingredient, rotigotine, or to one of its excipients
* Known allergy to sulphites
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection, or guardianship or curatorship.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of rotigotine administered at a dose of 4 mg/24h for 24 months in patients with ADPKD | throught 24 months
  Safety is defined by the occurrence of adverse events (AvE) and the occurrence of serious adverse events (SvA) for 24 months. The main safety criterion is based on the proportion of participants who experienced at least one EvIG during the 24 months of study follow-up such as the occurrence of serious reactions at the application site or certain behavioral disorders.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039